CLINICAL TRIAL: NCT04724629
Title: Prospective-randomized Adaptive Study, With Active Control to Evaluate the Efficacy and Safety of Interleukin (IL)-17 Inhibitor Treatment Versus Low Doses of IL-2 Versus Indirect IL-6 Inhibitor in Hospitalized Patients With Severe Forms of COVID-19
Brief Title: Survival TRial Using CytoKines in COVID-19 (STRUCK Trial)
Acronym: STRUCK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Science Valley Research Institute (Other)
Responsible Party: Principal Investigator, Fernando Bellissimo-Rodrigues, MD, PhD, Associated Professor - Dept of Social Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402422/2020-1
Record Dates: First submitted 2020-10-05; First posted 2021-01-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Covid19
Keywords: Colchicine; Ixekizumab; Cytokine storm; Lung vasculitis; Recombinant Human Interleukin-2
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — ixekizumab; aldesleukin; Colchicine; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multicenter, adaptive, open-label, randomized study design (1: 1: 1: 1 ratio), with an active comparator, superiority study, in severe to critical COVID19 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- IL-17 inhibitor (Ixekizumab) (Experimental): Patients will receive study medication Ixekizumab 80 mg per week, (SC) once a week for 4 weeks or until discharge.
  Interventions: Biological: Ixekizumab
- IL-2 (Aldesleukin) (Experimental): 1.5 million IU per day (SC) for 7 days or until discharge. Patients will receive study medication Aldesleukin 1.5 million IU per day (SC), for 7 days or until discharge.
  Interventions: Biological: Aldesleukin
- Indirect IL-6 inhibitor (Colchicine) (Experimental): Patients will receive study medication colchicine 0.5 mg every 8 hours for 3 days (PO), followed by 4 weeks (+/-7 days) 0.5 mg twice daily. If a dose is missed, it should not be replaced.
  Interventions: Drug: Colchicine
- Standard of care (Active Comparator): Standard treatment, supplementation of O2 ventilation + standard treatment of the institution, which may include Dexamethasone according to the institutional protocol.
  Interventions: Drug: Standard of care (SOC)

INTERVENTIONS:
Biological: Ixekizumab — 80 mg of IL-17 inhibitor
  Other Names: Taltz
  Arms: IL-17 inhibitor (Ixekizumab)
Biological: Aldesleukin — 1.5 million IU (low-dose) of IL-2
  Other Names: Proleukin
  Arms: IL-2 (Aldesleukin)
Drug: Colchicine — 0.5 mg of indirect IL-6 inhibitor
  Arms: Indirect IL-6 inhibitor (Colchicine)
Drug: Standard of care (SOC) — Active comparator (Corticoids and antiretrovirals)
  Arms: Standard of care

SUMMARY:
Currently, there are few approved treatments for COVID-19, antiretroviral (remdesivir) and corticoids. With about 15% of COVID-19 patients suffering from severe disease health system will be overwhelmed. Treatments approaches to inhibit viral replication (antiretroviral and extended spectrum antiviral drugs), such as Remdesivir and Hydroxychloroquine are being used. In severe cases, by CT scans investigators are able to observe that these patients seem to be dying with fibrosis and lung vasculitis. It is hypothesised that targeting vasculitis and lung inflammation secondary to the viral infection may help patients' survival (reducing mortality) and/or decrease time in mechanical ventilators. It is proposed a 4-arm trial, converted to 2 after interim analysis (60 patients for the initial phase, sample size recalculation after initial analysis and 2 arms beyond). In initial phase, IL-6 indirect inhibitor (colchicine), in first arm; IL-17 inhibitor, an innovative target never tested (at this moment) in COVID-19 severe patients, in second study arm. Both approaches (indirect IL-6 and Il-17) are related to modulation of inflammatory immune response. Finally, in third arm, IL-2 low dose. This cytokine was identified as Treg upregulation. Treg levels decrease in hepatitis C virus (HCV) associated vasculitis and increase in vasculitis resolution. In fourth arm, control group, standard of care. Initially, for the first 60 included patients, the study will comprise 4 arms (15 patients per arm, randomization ratio 1:1:1:1). An interim effectiveness and safety analysis at this point will guide the selection of one single treatment strategy (adaptative study) to be carried on after that, comparatively with the control group. The multi-site trial planned enrollment duration of 4-6 months and for each participant will be approximately 4 weeks. This trial will bring complementary data to the global effort in COVID-19 cases resolution.

ELIGIBILITY:
Inclusion Criteria:

* Positive result in the quantitative real-time PCR (qPCR) test for SARS-CoV-2 in the respiratory tract;
* Pneumonia confirmed by chest imaging and

  1. Respiratory rate ≥ 24 IRPM (for adults) or
  2. O2 saturation <93% or
  3. No improvement in O2 saturation, despite oxygen supply or
  4. Arterial hypotension; or
  5. Changes in capillary filling time; or
  6. Changes in the level of consciousness; or
  7. Oliguria;

IMPORTANT: The presence of increased respiratory rate or desaturation (items "a" and "b") are criteria for hospital admission. Items "c" to "g" are considered criteria for ICU admission

Following the recommendations of The São Paulo State Health Secretariat, resolution SS-28 of 03-Mar-2020, prepared by the Hospital das Clínicas of Medical School-USP.

Exclusion Criteria:

* Age <18 years;
* Refuse to sign the Informed Consent Form;
* Patient's decision that their involvement is not in their interest;
* Severe known liver disease (eg cirrhosis, with aminotransferase levels> 5 times the reference value limit);
* Pregnancy or breastfeeding period;
* Severe bacterial infection;
* Severe diarrhea;
* Diverticulitis or intestinal perforation;
* Infection known as HIV;
* Presence of one of the following uncontrolled or unstable cardiovascular diseases: stroke, ECG confirmed acute ischemia or myocardial infarction and / or clinically significant dysrhythmia; • Known history of gastrointestinal bleeding, uncontrolled peptic ulcer or uncontrolled duodenal ulcer;
* Known history of hemophilia or other bleeding disorders;
* History of organ transplantation, congenital immunodeficiency;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Ordinal scale of seven World Health Organization (WHO) categories of IL-17 inhibitor versus low dose IL-2 versus indirect IL-6 inhibitor (colchicine) versus standard treatment in the treatment of severe COVID-19 | On the 21st day of study, since inclusion.
  proportion of patients with clinical improvement, defined by an increase of two points in the ordinal scale of seven WHO categories

SECONDARY OUTCOMES:
Time until independence from oxygen therapy in days | During the follow-up period (30 days (+/- 2))
Ventilator free days (in days) | During the follow-up period (30 days (+/- 2))
Assessment of worsening pulmonary involvement, defined as the presence of one of these criteria (absence or presence) | At some point in Day 7, Day 14 and Day 28
  Need to increase the inspired fraction of O2 (FIO2) to keep oxygen saturation stable or the need for mechanical ventilation; b. Increase in the number and / or extension of affected lung areas on chest computed tomography.
In patients who needed mechanical ventilation, time to indicate mechanical ventilation | Day 0 up to 45 days
  (calculated in days, from entry into the protocol until orotracheal intubation, up to 45 days)
Duration of hospitalization, in survivors | On day 28
  In days
Analysis of in-hospital mortality | Day 0 up to 45 days
Analysis of general mortality | During the follow-up period (30 days (+/- 2))

OTHER OUTCOMES:
Correlation among the inflammatory proteins D-dimer, C- reactive protein (CRP), Lactate Dehydrogenase (LDH) Test, and ferritin with: | During the follow-up period (30 days (+/- 2))
  7 points WHO original scale; b. Time until independence from oxygen therapy; c. Need for mechanical ventilation; d. Days free of mechanical ventilation; e. Mortality
Changes from baseline of cytokine storm surrogate markers: white blood counts, lymphocyte counts, neutrophils counts, C-Reactive protein (CRP), ferritin (if applicable), D-dimer (if applicable) | at Day 0, Day 2, Day 4, Day 7, Day 14, Day 21 and Day 28 after randomization;
  Changes from baseline of cytokine storm surrogate markers: white blood counts, lymphocyte counts, neutrophils counts, CRP, ferritin (if applicable), D-dimer (if applicable)
Change in Score for Sepsis (SOFA score) | On days 7 and 14 of randomization
Analysis of secondary infections | During the follow-up period (30 days (+/- 2))
Qualitative and quantitative assessment of treatment- related adverse effects assessed by the Common Terminology Criteria for Adverse Event (CTCAE) version 5.0. | Within the first month

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rodrigues, MD, PhD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, USP, SP, Brazil; Eduardo Ramacciotti, MD, PhD, Study Chair — Hospital e Maternidade Dr. Christóvão da Gama, Grupo Leforte, Santo André, SP, Brazil; Leandro B Agati, PhD, Study Director — Hospital Leforte Liberdade, SP, Brazil; Esper Kallas, MD, PhD, Study Chair — Hospital das Clinicas de Sao Paulo (USP); Renato D Lopes, MD, PhD, Study Chair — Duke University
Locations (2):
- Brazil (2):
  - Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Hospital e Maternidade Christovão da Gama, Santo André, São Paulo